CLINICAL TRIAL: NCT02285283
Title: Randomized Double-Blinded Controlled Trial of Oral Antifungal for the Treatment of Fungal Sensitive Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Itraconazole for Fungal Sensitive Chronic Rhinosinusitis With Nasal Polyps
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment failure.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Amber Luong, Associated Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-14-0165
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Chronic Rhinosinusitis
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 capsules by mouth twice a day for 24 weeks
  Interventions: Drug: Placebo
- Itraconazole (Active Comparator): Two 100mg capsules by mouth twice a day for 24 weeks
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole
  Arms: Itraconazole
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this randomized controlled double-blinded trial is to determine if the addition of an oral antifungal to typical post-operative medical therapy can prevent or reduce the incidence of recurrence of nasal polyps in fungal sensitive patients with chronic rhinosinusitis with nasal polyps (CRSwNP).

DETAILED DESCRIPTION:
CRSwNP patients scheduled for medically-indicated sinus surgery will undergo screening ELIspot assay to identify patients with fungal sensitivity based on positive fungal induced interleukin 4 (IL-4) ELIspot. Enrolled fungal sensitive CRSwNP patients will undergo their sinus surgery and randomized into either placebo or itraconazole 200 mg taken by mouth twice a day (PO BID) for 24 weeks in addition to standardized post-surgical regimen (9 days of perioperative prednisone, saline irrigations and pain medication as needed). Patients will be followed as outpatient in rhinology clinic for 48 weeks total. During these post-op visits, compliance with medications will be determined. Patients will be questioned about any possible side effects or adverse events to post-operative medications. Then, the patients will be evaluated by 2 nasal specific quality of life questionnaires and nasal endoscopy. The goals of the nasal endoscopy are to evaluate the state of the sinus mucosa and to determine recurrence of nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for diagnosis of CRS with nasal polyps undergoing medically indicated sinus surgery

Exclusion Criteria:

* cystic fibrosis
* aspirin exacerbated respiratory disease
* uncontrolled or unstable chronic diseases such as uncontrolled diabetes
* active or history of cancer
* HIV positive
* history of liver or kidney disease
* history of disease with effects on immune system
* pregnant
* allergy to triazole antifungals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Luong, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Medical School at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 2 capsules by mouth twice a day for 24 weeks
  Placebo
- Itraconazole: Two 100mg capsules by mouth twice a day for 24 weeks
  Itraconazole
Period: Overall Study
Arm/Group | Placebo | Itraconazole
Started | 29 | 29
Completed | 25 | 20
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Itraconazole | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 28 | 25 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 22 | 17 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Nasal Polyps Requiring Intervention
Description: Recurrence of nasal polyps requiring intervention
Time Frame: 48 weeks
Population: 33 participants were lost to follow up, and data was not collected for these 33 participants (16 in the placebo arm and 17 in the itraconazole arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Itraconazole
Number analyzed (Participants) | 13 | 12
Participants | 3 | 4

2. Secondary Outcome: Number of Participants With Adverse Events During Time Frame of Taking Medication/Placebo
Description: Adverse events during time frame of taking medication/placebo
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Itraconazole
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: 33 participants were lost to follow up, and data was not collected for these 33 participants (16 in the placebo arm and 17 in the itraconazole arm).
Arm/Group | Placebo | Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT02285283/Prot_SAP_000.pdf